CLINICAL TRIAL: NCT06204965
Title: The Impact of Time-restricted Eating on the Composition of the Intestinal Microbiota and Metabolic and Neurohormonal Parameters of Women With Polycystic Ovary Syndrome
Brief Title: The Impact of Time-restricted Eating on the Outcomes Associated With Polycystic Ovary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Joanna Bajerska (Other)
Responsible Party: Sponsor-Investigator, Joanna Bajerska, Associate Professor, Poznan University of Life Sciences
Organization: Poznan University of Life Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 646/23
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Intermittent Fasting; Microbiota; Neurotransmitter Agents; Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: Women with Polycystic Ovary Syndrome (n=52), aged 18-40.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted eating group (TRE group) (Experimental): Participants assigned to the TRE group will be instructed to continue eating their usual diet during the experiment (without any qualitative or quantitative restrictions), but to eat it within a limited time frame - from 9:00 a.m. to 5:00 p.m., and then fast until the next day ( protocol 8/16).
  Interventions: Behavioral: Time-restricted eating
- Non-fasting group (No Intervention): Participants assigned to the control group will receive only dietary recommendations consistent with the healthy eating plate. Additionally, the recommended energy intake will be individually determined for each patient using the PPM (calculated using the Harris-Benedict formula) multiplied by the physical activity factor.

INTERVENTIONS:
Behavioral: Time-restricted eating — Time-restricted eating (TRE) is a dietary pattern where food intake is restricted to 8 hours of the day with no limitation on nutrient quality or quantity. Participants assigned to the intervention group will eat their usual diet from 9:00 a.m. to 5:00 p.m., and then fast until the next day (protocol 8/16). During the 16-hour fast, only hot and cold drinks will be allowed, i.e. coffee, tea or tea and water, but all products and dishes with energy value (including coffee cream, sweet teas, alcohol, snacks, etc.) will be prohibited. The TRE protocol will be implemented 7 days a week for a period of 3 months (12 weeks).
  Arms: Time-restricted eating group (TRE group)

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is a disorder that affects approximately 10-15% of women of reproductive age. Increased activity of the hypothalamic-pituitary-ovarian (HPO) axis is considered to be one of the main factors associated with the pathogenesis of PCOS. The regulation of the activity of this axis is influenced by the following factors: insulin resistance and the activity of kisspeptins in the hypothalamus. It is suggested that intestinal dysbiosis may also play a key role in the pathogenesis of PCOS. It was noticed that the presence of bacteria producing gamma-aminobutyric acid in the intestine is positively correlated with the concentration of luteinizing hormone (LH) in the serum, which indicates the relationship between the functioning of the gut-brain axis and PCOS. A dysbiotic factor is an incorrect diet and inappropriate timing of its consumption, which may also lead to inhibition of kisspeptin expression in the hypothalamus and cause menstrual disorders.

Due to the fact that most obese women with PCOS eat significantly more meals in the second part of the day, and these meals are characterized by a significant supply of fat and simple sugars, intestinal dysbiosis seems to be an important cause of the observed disorders, while the use of chrononutrition, consisting in synchronizing meal times with endogenous 24-hour circadian rhythms may partially restore eubiosis in the intestine and improve the reproductive, metabolic and neurohormonal health of women with PCOS. Time-restricted feeding (TRF), which involves eating food usually within 8 hours followed by 16 hours of fasting, seems to be a regime that allows restoring eubiosis in the intestinal microbiota and improving the quality of life of women with PCOS. So far, only one study has been conducted among women with PCOS who used TRF for 5 weeks and a number of positive changes were demonstrated (hormonal or metabolic). However, this study did not include an assessment of the microbial and neurohormonal parameters, which seems to be a key issue.

Taking the above into account, it was hypothesized that TRF may be an appropriate therapeutic tool for women with PCOS, which will positively affect metabolic and hormonal parameters by changing the composition of the intestinal microbiota. Therefore, the main aim of the experiment is to investigate the impact of TRF on the composition of the intestinal microbiota, its metabolites, and metabolic and neurohormonal parameters in women with PCOS.

DETAILED DESCRIPTION:
Fifty two women, aged 18-40, will be recruited for the study. The investigators calculated the sample size using G*Power software (RRID:SCR_013726); the sample size of the participants was also determined. The effect size was calculated to be 1.04 on the basis of the differences in body fat mass between baseline values and values after 6-weeks of application of time-restricted eating by PCOS women. With an alpha value of 0.05, a sample size of eight mice per group would yield a power of 0.95.

Women recruited for the study will be provided with detailed information regarding: the purpose of the study, the study protocol, the measurements performed and the duration of the study. Recruitment will take place via social networking sites, i.e. Facebook, where target groups will be found, bringing together women with PCOS, and posts with an announcement and a contact form will be placed there. After obtaining consent to participate in the study, a group of qualified women will undergo a general medical interview by Jakub Noskiewicz, Ph.D., which will include a personal interview, including current medications and supplements taken, medical history and a basic physical examination - examination, percussion. If the interview reveals an existing infection, a chronic disease in the acute phase, a suspicion of e.g. anemia, infectious skin diseases or malnutrition, or the intake of medications constituting an exclusion criterion, the patient will not be qualified for the study. During this interview, participants will be asked to provide medical documentation confirming they suffer from PCOS.

Participants will be randomly assigned (using a specialized program) to two groups - control and intervention. Research participants assigned to the control group will receive dietary recommendations consistent with the healthy eating plate. Additionally, the recommended daily energy intake will be individually determined for each patient. Participants assigned to the TRF group will be instructed to continue eating their usual diet during the experiment (without any qualitative or quantitative restrictions), but to eat it within a limited time frame - from 9:00 a.m. to 5:00 p.m., and then fast until the next day ( protocol 8/16). The duration of the study will be 3 months (12 weeks).

A nutritional assessment of the diet will be carried out (KomPAN questionnaire). The nutritional assessment will be additionally supplemented by an interview from the last 24 hours. Then, the recruited women will be randomly assigned to the intervention group, using time-restricted nutrition, or the control group, using the principles of the healthy eating plate. The duration of the experiment will be 12 weeks, with follow-up visits scheduled at 4-week intervals. At the beginning of the experiment and at follow-up visits, women will have blood drawn (per 18 ml) to assess biochemical parameters. Each time, a stool sample will also be collected to assess the composition of the intestinal microbiota and short-chain fatty acids, and an analysis of body composition, bone density and anthropometric parameters will be carried out. During the last visit in week 12, women will be asked to fill out the KomPAN questionnaire again, which will be supplemented by an interview from the last 24 hours. Each time, an interview will be conducted regarding the women's well-being and adherence to the recommendations provided. The level of adherence to the eating window will be verified using a diary in which women will write down each day when they ate their first and last meals.

The following specific analyses are planned:

* Assessment of anthropometric parameters (body weight, height, waist circumference, hip circumference) as well as body composition and bone density.
* Assessment of carbohydrate metabolism parameters (concentration of glucose, insulin, calculation of HOMA-IR, HOMA-β, QUICKI), lipid metabolism (concentration of total cholesterol (T-C), LDL cholesterol (LDL-C), HDL cholesterol (HDL-C) , non-HDL cholesterol (non-HDL-C) and triglycerides)
* Assessment of hormonal parameters (FSH, LH, testosterone, SHBG) and lipopolysaccharide in the blood.
* Assessment of neurohormonal parameters (kisspeptin, gamma-aminobutyric acid) in the blood.
* Assessment of the composition of intestinal microbiota and short-chain fatty acids in women's feces.

Normality of the obtained data distribution will be tested using the Shapiro-Wilk test. The Kruskal-Wallis test then will be used for nonnormally distributed data and the Tukey HSD test will be used for normally distributed data. A p value of less than 0.05 was considered statistically. The microbiota composition will be analyzed using RStudio (R version 4.0.3 (2020-10-10)) with packages including phyloseq, microbiome, and vegan. Taxa will be filtered by removing all those not assigned to any phylum. Only taxa with abundances over 0.25% in at least one sample will left in the dataset. All analyses of gut microbiota composition will be performed on the basis of the relative abundances (RA) of the OTUs.

The data collected in the planned studies will include the results of measurements and their statistical analyzes. All data will be collected directly by team members and coded. Detailed instructions on data collection will be prepared by the team leader and each member will need to read and receive appropriate training. All biochemical and anthropometric measurements will be performed in at least two repetitions and will be checked by another team member. All used specialized equipment will be properly calibrated before each use (scale, body composition analyzer, Nanodrop spectrophotometer).

ELIGIBILITY:
Inclusion criteria

* Age 18-40
* suffering from Polycystic Ovary Syndrome, confirmed by appropriate medical documentation
* BMI >25 kg^m2

Exclusion criteria

* Taking medications regulating carbohydrate, lipid as well as medications affecting body weight in the last 3 months (will be assessed during a general medical interview conducted by Jakub Noskiewicz, MD, PhD)
* Taking antibiotics in the last 3 months
* Smoking in the last 3 months and alcohol consumption >100 g per week
* Competitive sports practice
* Significant body weight fluctuations in the 3 months before the start of the study (>5%)
* Pregnant or breastfeeding women
* BMI <25 kg^m2

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | Week 0 (pre-intervention), week 4, week 8 and week 12 (post-intervention)
  Body weight measurement in a standing position, without shoes, in light clothing, on an electronic scale with an accuracy of 0.1 kg.
Change in circumferences | Week 0 (pre-intervention), week 4, week 8 and week 12 (post-intervention)
  Waist and hip measurements will be taken using an elastic tape. Waist circumference measurement - the tape is placed horizontally or slightly obliquely halfway between the lower edge of the ribs and the upper crest of the ilium. Measurement performed during apnea.
Change in body composition | Week 0 (pre-intervention), week 4, week 8 and week 12 (post-intervention)
  Body composition will be measured using dual-energy X-ray absorptiometry (DXA) as a method that uses the phenomenon of weakening the beam of ionizing radiation passing through tissues of various densities. This method is safe and non-invasive. The mass of adipose tissue, including visceral fat tissue, the mass of lean tissue are measured (expressed in the same unit - kilograms)
Change in composition of the intestinal microbiota | Week 0 (pre-intervention), week 4, week 8 and week 12 (post-intervention)
  Participants will be asked to provide stool samples at each scheduled meeting. Detailed instructions on sample collection and transport will be provided by the people conducting the study, and participants will receive containers containing preservative liquid. Bacterial DNA will be isolated from the provided stool samples using the QIAmp Fast DNA Stool Mini Kit. Then, the DNA will be properly secured and sent to an external company, Genomed S.A. (Warsaw, Poland), in which the assessment of microbiota will be carried out by metagenomic 16s rRNA sequencing using the V3-V4 region. Then, a bioinformatics analysis will be performed in the R environment using packages such as phyloseq, vegan, microbiome.
Change in selected hormonal parameters | Week 0 (pre-intervention), week 4, week 8 and week 12 (post-intervention)
  Blood will be collected four times from the antecubital vein on an empty stomach, into test tubes with clotting granules (a single sample will amount to a total of 18 ml). The serum will be obtained by centrifugation of a venous blood clot. Hormonal parameters (FSH, LH, testosterone, SHBG), will be performed using the ELISA enzyme-linked immunosorbent assay (expressed in the same unit - pg/ml)
Change in lipid profile | Week 0 (pre-intervention), week 4, week 8 and week 12 (post-intervention)
  Blood will be collected four times from the antecubital vein on an empty stomach, into test tubes with clotting granules (a single sample will amount to a total of 18 ml). The serum will be obtained by centrifugation of a venous blood clot. Total cholesterol (T-C), low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C) and triglycerides concentrations will be determined using the Thermo Scientific Konelab 20i automatic biochemical analyzer (enzymatic method ). The nonHDL-C parameter will be calculated using the formula: nonHDL-C = T-C - HDL-C (expressed in the same unit - mg/dl or mmol/l).
Change in glucose metabolism | Week 0 (pre-intervention), week 4, week 8 and week 12 (post-intervention)
  Blood will be collected four times from the antecubital vein on an empty stomach, into test tubes with clotting granules (a single sample will amount to a total of 18 ml). The serum will be obtained by centrifugation of a venous blood clot. Insulin concentration will be performed using the ELISA enzyme-linked immunosorbent assay, while glucose will be determined using the Thermo Scientific Konelab 20i automatic biochemical analyzer (enzymatic method ) (expressed in the same unit - mg/dl or mmol/l).

SECONDARY OUTCOMES:
Assessment of changes in eating behavior pre- and post-intervention | Week 0 (pre-intervention), week 4, week 8 and week 12 (post-intervention)
  Nutrition assessment will be carried out using the validated questionnaire for examining dietary views and habits for people aged 16 to 65 (KomPAN) questionnaire. The obtained data will be transformed from the rank assigned to consumption frequency categories from 1 - 6 to a daily frequency from 0-2. Diet quality indicators will be calculated - pro-Healthy-Diet-Index-10 (pHDI - range 0-20), non-Healthy-Diet-Index-14 (nHDI - range 0 - 28), Diet-Quality-Index (DQI - range -100-100). The higher the value of the pHDI or DQI index, the greater the intensity of nutritional features beneficial to health and the better the quality of the diet. The higher the value of the nHDI index, the greater the intensity of nutritional characteristics unfavorable for health and the worse the quality of the diet. In addition, an interview from the last 24 hours will be conducted.
Change in bone density | Week 0 (pre-intervention), week 4, week 8 and week 12 (post-intervention)
  Bone density will be measured using dual-energy X-ray absorptiometry (DXA) as a method that uses the phenomenon of weakening the beam of ionizing radiation passing through tissues of various densities. This method is safe and non-invasive.
Change in the concentration of short-chain fatty acids in feces | Week 0 (pre-intervention), week 4, week 8 and week 12 (post-intervention)
  Quantitative and qualitative determination of short-chain fatty acids in feces will be carried out using the gas chromatography method with flame ionization detection (GC-FID). The research will be carried out at the Department and Department of Bromatology, Medical University of Poznań.
Change in the expression of genes encoding kisspeptin and gamma-aminobutyric acid | Week 0 (pre-intervention), week 4, week 8 and week 12 (post-intervention)
  The expression of genes encoding kisspeptin (KISS1) and gamma-aminobutyric acid (GABA) will be assessed using the quantitative RT-PCR method using TaqMan oligonucleotide probes specific for these genes. All blood test determinations and gene expression will be performed using analyzers and devices that are part of the equipment of the Molecular Metabolism Research Laboratory. Biological and genetic material will be stored at -80°C for further research at the Department of Human Nutrition and Dietetics, Faculty of Food Sciences and Nutrition, University of Life Sciences in Poznań. Blood will be collected by a member of the research team, an active physician (specializing in surgery), PhD Jakub Noskiewicz.
Change in intestinal barrier integrity | Week 0 (pre-intervention), week 4, week 8 and week 12 (post-intervention)
  Blood will be collected four times from the antecubital vein on an empty stomach, into test tubes with clotting granules (a single sample will amount to a total of 18 ml). The serum will be obtained by centrifugation of a venous blood clot. Lipopolysaccharide concentrations will be assessed using the ELISA enzyme-linked immunosorbent assay.
Change in neurohormonal status | Week 0 (pre-intervention), week 4, week 8 and week 12 (post-intervention)
  Blood will be collected four times from the antecubital vein on an empty stomach, into test tubes with clotting granules (a single sample will amount to a total of 18 ml). The serum will be obtained by centrifugation of a venous blood clot. Kisspeptin and gamma-aminobutyric acid concentrations will be performed using the ELISA enzyme-linked immunosorbent assay.

CONTACTS AND LOCATIONS:
Overall Officials: Agata Chmurzyńska, Prof., Study Chair — Department of Human Nutrition and Dietetics, Poznań University of Life Sciences
Locations (1):
- Poznań University of Life Sciences, Poznan, Greater Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Numerical data, statistics and graphs data will be deposited in the Open Data Repository RepOD - the PULS institutional repository, and made publicly available in the Repository at the latest at the time when the publication presenting research data is published including a maximum 36-month embargo period due to the requirements and specifics of the publication of the article presenting the research results. Upon publication, the embargo will be lifted immediately.
  Unless there is a clear indication to the contrary, the data will be made available in the RepOD repository under a CC BY 4.0 license. Data not stored in RepOD will be stored long term as described in 3.1.
  Raw and processed data will be stored for at least 10 years. Personal data will be deleted after the pseudonymization process.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD data will be made available after publication of all planned articles presenting the results of the planned experiment for a period of 10 years.
Access Criteria: All persons having access to data have to be authorised to process personal data. A secured work e-mail is used for correspondence. Access to collected and processed sensitive data will be limited solely to the group of authorised users. The Head of the project authorises individuals to have access to data.
  The e-mail requesting access to the IPD should include your name and surname, academic degree and affiliation. Data will only be made available after the person's identity has been verified and the purpose of using the data is clear (e.g. meta-analysis). Then, the data owner will verify the need to have the data and send it in a password-protected form. All data will be pseudonymized.

REFERENCES:
- [Background] Li C, Xing C, Zhang J, Zhao H, Shi W, He B. Eight-hour time-restricted feeding improves endocrine and metabolic profiles in women with anovulatory polycystic ovary syndrome. J Transl Med. 2021 Apr 13;19(1):148. doi: 10.1186/s12967-021-02817-2. PMID 33849562
- [Background] Torres PJ, Ho BS, Arroyo P, Sau L, Chen A, Kelley ST, Thackray VG. Exposure to a Healthy Gut Microbiome Protects Against Reproductive and Metabolic Dysregulation in a PCOS Mouse Model. Endocrinology. 2019 May 1;160(5):1193-1204. doi: 10.1210/en.2019-00050. PMID 30924862
- [Background] Liao B, Qiao J, Pang Y. Central Regulation of PCOS: Abnormal Neuronal-Reproductive-Metabolic Circuits in PCOS Pathophysiology. Front Endocrinol (Lausanne). 2021 May 28;12:667422. doi: 10.3389/fendo.2021.667422. eCollection 2021. PMID 34122341
- [Background] Tremellen K, Pearce K. Dysbiosis of Gut Microbiota (DOGMA)--a novel theory for the development of Polycystic Ovarian Syndrome. Med Hypotheses. 2012 Jul;79(1):104-12. doi: 10.1016/j.mehy.2012.04.016. Epub 2012 Apr 27. PMID 22543078
- [Background] Minabe S, Iwata K, Tsuchida H, Tsukamura H, Ozawa H. Effect of diet-induced obesity on kisspeptin-neurokinin B-dynorphin A neurons in the arcuate nucleus and luteinizing hormone secretion in sex hormone-primed male and female rats. Peptides. 2021 Aug;142:170546. doi: 10.1016/j.peptides.2021.170546. Epub 2021 Mar 29. PMID 33794282